

## **Protocol ARO-011**

Pilot study of Crenolanib Combined with Standard Salvage Chemotherapy in Subjects with Relapsed/Refractory Acute Myeloid Leukemia

**IND Number: 118143** 

The information contained in this protocol is confidential and is intended for the use of clinical investigators. It is the property of AROG Pharmaceuticals, Inc., or its subsidiaries and should not be copied by or distributed to persons not involved in the clinical investigation of crenolanib besylate, unless such persons are bound by a confidentiality agreement with AROG Pharmaceuticals, Inc., or its subsidiaries.

Version Number: 3.0

Version Date: June 7, 2016

AROG Pharmaceuticals, Inc. 5420 LBJ Freeway, Suite 410 Dallas, TX 75240

# **TABLE OF CONTENTS**

| T | ABLE O | F CONTENTS | 0 |
|---|---|---|---|
| LI | ST OF | ABBREVIATIONS | 3 |
| D | EFINIT | ON OF TERMS | 5 |
| 1. | SYN | OPSIS | 6 |
| 2. | BAC | KGROUND AND STUDY RATIONALE | 11 |
| | 2.1 U | NMET MEDICAL NEED IN RELAPSED OR REFRACTORY ACUTE MYELOID LEUKEMIA | 11 |
| | | HYSICIAN'S CHOICE OF SALVAGE CHEMOTHERAPY AGENTS IN RELAPSED/REFRACTORY AML | |
| | | FICACY OF HAM, MEC AND FLAG-IDA IN RELAPSED/REFRACTORY AML | |
| | 2.4 Cı | INICAL EVIDENCE OF COMBINING A TYROSINE KINASE INHIBITOR WITH CHEMOTHERAPY IN AML PATIENTS | 13 |
| | | T3 LIGAND LEVELS INCREASE FOLLOWING ADMINISTRATION OF CHEMOTHERAPY | |
| | | VERVIEW OF CRENOLANIB | |
| | 2.7 RA | ATIONALE FOR COMBINING CRENOLANIB WITH HAM, MEC, OR FLAG-IDA | 16 |
| 3. | STU | DY OBJECTIVES | 16 |
| | 3.1 PF | RIMARY OBJECTIVE | 16 |
| | 3.2 SE | CONDARY OBJECTIVES | 16 |
| 4. | STU | DY DESIGN | 17 |
| | 4.1 Es | TIMATED STUDY DURATION | 17 |
| 5. | STU | DY POPULATION | 18 |
| | 5.1 IN | CLUSION CRITERIA | 18 |
| | | CLUSION CRITERIA | |
| | 5.3 Sc | REENING FAILURES | 20 |
| 6. | ASS | ESSMENTS & SCHEDULE | 20 |
| | 6.1 Sc | REENING ASSESSMENTS | 20 |
| | 6.2 O | N-STUDY BASELINE ASSESSMENTS | 21 |
| | | ALUATION DURING TREATMENT | |
| | | ALUATION DURING FOLLOW-UP | |
| | | ND OF STUDY AND POST-TREATMENT FOLLOW-UP VISITS | |
| | 6.6 ST | 'UDY CALENDAR | 24 |
| 7. | STU | DY TREATMENT | 25 |
| | 7.1 O | VERVIEW OF STUDY TREATMENT: INVESTIGATIONAL PRODUCT, CRENOLANIB | 25 |
| | 7.2 CF | RENOLANIB DOSE LEVELS AND DOSE ADJUSTMENTS | 26 |
| | | OSE-LIMITING TOXICITY | |
| | | UDY TREATMENT MANAGEMENT | |
| | 7.4.1 | | |
| | 7.4.2 | | |
| | 7.4.3 | | |
| | 7.4.4<br>7.4.5 | · | |
| | 7.4.5<br>7.4.6 | | |
| | | DIVIDING DIVIDING STATES OF THE STATES OF TH | |
| 8. | | CONTINUATION | |
| -• | | | |
| | | UDY TREATMENT DISCONTINUATION AND PREMATURE WITHDRAWAL | |
| | 0.2 31 | ODI DISCONTINUATION | 33 |

# Protocol ARO-011

| Version 3 | 3.0 | June 7, 2016 |
|---|---|---|
| 8.3 | SITE DISCONTINUATION | 33 |
| 9. CO | ORRELATIVE STUDIES | 34 |
| 9.1 | PERIPHERAL BLOOD FOR PHARMACOKINETIC ASSAY | 34 |
| 10. CI | RITERIA FOR RESPONSE | 36 |
| 10.1 | Response Criteria | 36 |
| 11. AI | DVERSE EVENT REPORTING | 37 |
| 11.1 | Definitions | 37 |
| 11.2 | DETERMINATION OF SEVERITY | 38 |
| 11.3 | DETERMINATION OF RELATEDNESS | 38 |
| 11.4 | REPORTING OF ADVERSE EVENTS | 38 |
| 11.5 | REPORTING OF SERIOUS ADVERSE EVENTS | 39 |
| 11.6 | Pregnancy | 41 |
| 12. ST | TATISTICAL CONSIDERATIONS | 42 |
| 12.1 | STATISTICAL AND ANALYTICAL PLANS | 42 |
| 12 | 2.1.1 General considerations | 42 |
| 12 | 2.1.2 Determination of sample size | 42 |
| 12.2 | SAFETY MONITORING AND STOPPING RULES FOR THE STUDY | 42 |
| 13. DA | ATA QUALITY MANAGEMENT | 44 |
| 13.1 | Data Safety Monitoring Plan | 44 |
| 13.2 | Data Quality Assurance | |
| 14. RI | EFERENCES | 45 |
| 15. AI | PPENDIX I, ADMINISTRATIVE PROCEDURES | 49 |
| 16. AI | PPENDIX II, PATIENT DIARIES: CRENOLANIB | 52 |
| 17. AI | PPENDIX III. LABORATORY MANUAL | 55 |
| 17.1 | FORM 1 ARO-011 INDUCTION 1 DAY PHARMACOKINETICS DATA COLLECTION FORM | |
| 17.2 | FORM 2 ARO-011 INDUCTION 1 DAY PHARMACOKINETICS DATA COLLECTION FORM | |
| | PPENDIX IV. CONTACT INFORMATION | |
| 19. AI | PPENDIX V. HY'S LAW | 62 |
| | PPENDIX VI. CYP3A4 DRUGS POTENTIALLY AFFECTING CRENOLANIB | |
| PHARM | AACOKINETICS | 66 |

| List | of | Fig | gur | es |
|------|----|-----|-----|----|
|------|----|-----|-----|----|

| Figure 1 Overall survival estimates in the intention-to-treat population of elacytarabine versu | |
|---|---|
| investigator's choice of current salvage therapies by Kaplan-Meier test | 11 |
| Figure 2 Overall survival in the intention-to-treat population of investigator's choice of curre | ent |
| salvage therapies by Kaplan-Meier test | 12 |
| Figure 3 Event-free survival in the sorafenib arm vs. placebo | 14 |
| Figure 4 FLT3 ligand levels increase following multiple regimens of intensive chemotherapy | y 14 |
| Figure 5 Peripheral blast clearance in FLT3 mutant AML patients treated with crenolanib | 15 |
| List of Tables | |
| Table 1 30-day, 60-day mortality rates of elacytarabine and investigator's choice | 11 |
| Table 2 Pivotal studies using the HAM regimen as salvage | 13 |
| Table 3 Screening Assessments | |
| Table 4 On-Study Baseline Assessments | 21 |
| Table 5 Post-treatment Discontinuation Visit Assessments | 22 |
| Table 6 Crenolanib dose reduction schedule | |
| Table 7 Crenolanib dose reduction for non-hematologic toxicities related to crenolanib | 26 |
| Table 8 Crenolanib dose reduction for bilirubin elevation | |
| Table 9 Crenolanib dose reduction for elevation of AST, ALT, Alk Phos | |
| Table 10 Suggested therapy for nausea and vomiting (ASCO 2011 guidelines [41]) | |
| Table 11 Suggested therapy for diarrhea | |

# LIST OF ABBREVIATIONS

Term Definition
AE Adverse Event

ALT Alanine aminotransferase
AML Acute myeloid leukemia
AST Aspartate aminotransferase

AUC Area under the curve

BID Twice daily

CBC Complete blood count

C<sub>max</sub> Maximum concentration of drug in serum

CMP Complete metabolic panel

CR Complete remission

CRi Complete remission with incomplete count recovery

CRF Case report form

CTCAE Common terminology criteria for adverse events

DARF Drug accountability record form

DLT Dose limiting toxicity
DOR Duration of response
EC Ethics Committee

ECOG Eastern Cooperative Oncology Group

eCRF Electronic case report form

EFS Event-free survival EKG Electrocardiogram

EOS End of study

FLAG Fludarabine, Ara-C, G-CSF FLT3 FMS-like tyrosine kinase 3

FLT3-ITD FMS-like tyrosine kinase 3 – internal tandem duplication

FLT3-TKD FMS-like tyrosine kinase 3 – tyrosine kinase domain

GCP Good clinical practice
GVHD Graft versus host disease

HAM High-dose cytarabine and mitoxantrone

HiDAC High-dose cytarabine

HR Hazard ratio

HSCT Hematopoietic stem-cell transplant

IB Investigator Brochure

Protocol ARO-011

Version 3.0 June 7, 2016

ICF Informed consent form

ICH International Conference on Harmonisation

Ida Idarubicin

IDAC Intermediate-dose cytarabine

IMP Investigational medicinal product(s)

IRB/IEC Institutional review board/ Independent ethics committee

ITT Intent-to-treat

IVRS Interactive voice response system

KM curve Kaplan-Meier curve LFT Liver function test

MEC Mitoxantrone, Etoposide, Cytarabine

MTD Maximum tolerated dose

MTZ Mitoxantrone

ORR Overall response rate

OS Overall survival
PD Progressive disease

PDGFR $\alpha$  Platelet-derived growth factor receptor alpha

PFS Progression-free survival

PK Pharmacokinetic
PR Partial response
PS Performance Status

RECIST Response Evaluation Criteria In Solid Tumors

RFS Relapse-free survival R/R Relapsed/Refractory

RR Response Rate

RTK Receptor tyrosine kinase SAE Serious adverse event

SD Stable disease SOC Standard of care

SUSAR Suspected Unexpected Serious Adverse Reactions

 $t_{1/2}$  Half-life

TID Three times daily

TKI Tyrosine kinase inhibitor

t<sub>max</sub> Time that drug is at maximum concentration in serum

QD Once daily

Upper limit of normal ULN

Women of child-bearing potential **WOCBP** 

# **DEFINITION OF TERMS**

| 1 erm | Definition |
|---|---|
| Adverse Drug | Any adverse event that is deemed to be at least possibly related to the study |
| Reaction | drug. |
| | A |

| Adverse Drug | Any adverse event that is deemed to be at least possibly related to the study |
|---|---|
| Reaction | drug. |
| Audit | A systematic and independent examination of the trial-related activities and documents to determine whether the evaluated trial-related activities were conducted, and the data were recorded, analyzed, and accurately reported according to the protocol, applicable standard operating procedures (SOPs), good clinical practice (GCP), and the applicable regulatory requirement(s). |
| Case Report Form (CRF) | Sometimes referred to as clinical report form: a printed or electronic form for recording study participants' data during a clinical study, as required by the protocol. |
| Compliance | Adherence to all the trial-related requirements, good clinical practice (GCP) requirements, and the applicable regulatory requirements. |
| Consent | The act of obtaining informed consent for participation in a clinical trial from subjects deemed eligible or potentially eligible to participate in the clinical trial. Individuals entered into a trial are those who sign the informed consent document directly or through their legally acceptable representatives. |
| Enrolled Subject | An enrolled subject is a subject who has signed the informed consent form, completed all screening evaluations, has been deemed eligible for the trial by the investigator and sponsor and has been enrolled. |
| Ethics Committee | All appropriate properly constituted committees or boards recognized by the appropriate regulatory agencies for approving clinical studies. Including the independent ethics committee and institutional review boards. |
| Investigator | A person responsible for the conduct of the clinical trial at a trial site. If a trial is conducted by a team of individuals at a trial site, the investigator is the responsible leader of the team and may be called the principal investigator. |
| Institutional Review<br>Board/ Ethics Review<br>Board (IRB/ERB) | A board or committee (institutional, regional, or national) composed of medical and nonmedical members whose responsibility is to verify that the safety, welfare, and human rights of the subjects participating in a clinical trial are protected. |
| Regulation | All appropriate regulations, laws and guidelines. |
| Screening Period | The screening period begins when the subject signs the Informed Consent Form and continues until randomization. |
| Screen Failure | A screen failure refers to subjects who have signed the Informed Consent Form but do not subsequently enroll in the trial. Data from these subjects will be recorded in the screening log, but not entered into the study database. |
| Treatment period | The time period from administration of the first dose of study drug through the end of the one month post-treatment discontinuation visit. |

## 1. SYNOPSIS

## Name of Investigational Product

Crenolanib Besylate

# **Title of Study**

Pilot study of Crenolanib Combined with Standard Salvage Chemotherapy in Subjects with Relapsed/Refractory Acute Myeloid Leukemia

# **Version and Date of Protocol**

Version 3.0, June 7, 2016

# Planned number of subjects and investigational sites

Approximately 72 subjects (~24 in each cohort) will be enrolled across approximately 10 sites in the U.S.

# **Study Rationale**

Treatment of newly-diagnosed acute myeloid leukemia (AML) with standard chemotherapy regimens, such as anthracyclines and cytarabine, can lead to high complete remission (CR) rates (ranging from 60-70%). Unfortunately, the majority of these patients will relapse.

Upon relapse, the prognosis for a second remission or response in these patients significantly worsens. Currently, patients who are refractory or relapsed following standard induction therapy have no standardized treatment options. Several combinations have been suggested and each achieve similar outcome. High-dose cytarabine combined with mitoxantrone (HAM) has been shown to be associated with high CR rates in relapsed/refractory (R/R) AML. Two additional aggressive salvage chemotherapies, as per National Comprehensive Cancer Network (NCCN) guidelines, are also common options for relapsed/refractory patients: the combination of mitoxantrone, etoposide, and cytarabine (MEC) and the combination of fludarabine, cytarabine, G-CSF and idarubicin (FLAG-Ida). However, it has been proven difficult to achieve full prolonged responses with these chemotherapy agents alone.

Recent studies have shown that in AML, the addition of a tyrosine-kinase inhibitor (TKI) to standard chemotherapy in a sequential manner is feasible and associated with anti-leukemic efficacy. A randomized study (SORAML) has shown that the addition of a sorafenib to standard chemotherapy resulted in a significantly prolonged event-free survival (EFS) and relapse-free survival (RFS). This data has also suggested that this treatment regimen can be beneficial and effective in both FLT3 (Fms-related tyrosine kinase 3) wild-type and FLT3 ITD (FLT3 – Internal Tandem Duplication) AML.

Crenolanib besylate is a second generation TKI with high potency and selectivity against both wild-type FLT3 and its constitutively active mutant isoforms including FLT3-ITD mutation and also tyrosine kinase domain (TKD) point mutations including the D835 TKD mutation. Clinical safety data of crenolanib is available for over 200 patients. Specifically, there are data in 66 patients with R/R FLT3 ITD and/or TKD mutant AML, which demonstrates clinical benefit in approximately 50% of these AML patients with responses that included complete remission (CR), complete remission with incomplete blood count recovery (CRi) and partial remission (PR).

The proposed study is designed combine crenolanib with salvage chemotherapies, including HAM, MEC or FLAG-Ida to treat patients with R/R AML irrespective of FLT3 status. The rationale for this study is as follows:

- (1) There is clinical evidence for improved event-free survival in AML with the combination of a TKI and chemotherapy;
- (2) HAM, MEC, and FLAG-Ida have been shown to improve the outcome in patients with R/R AML;

(3) Sequential administration of chemotherapy followed by a TKI is feasible and can achieve synergistic cytotoxicity.

# **Study Design**

Open label, dose de-escalation, phase 1b pilot trial of crenolanib with standard salvage chemotherapy. Subjects may receive up to 2 cycles of induction with standard salvage chemotherapy followed by crenolanib. Each arm will enroll approximately 24 patients (72 total); stratification to each arm will be per physician's choice.



## Arm A (HAM + crenolanib)

Subjects 18-60 years of age who have not undergone a prior allogeneic hematopoietic stem cell transplant (HSCT):

| • | Mitoxantrone | 10 mg/m <sup>2</sup> IV, over ≤ 30 mins | days 1-3 |
|---|---|---|---|
| • | Cytarabine | 1000 mg/m <sup>2</sup> IV, over 3 hours | days 1-6 |
| • | Crenolanib | 100 mg TID p.o. | starting day 7 (+3 day) |

For subjects > 60 years, or subjects who have undergone a prior allogeneic HSCT, or subjects who need a second re-induction HAM cycle, the following reduced doses will be used:

| • | Mitoxantrone | $8 \text{ mg/m}^2 \text{ IV}$ , over $\leq 30 \text{ mins}$ | days 1-3 |
|---|---|---|---|
| • | Cytarabine | 500 mg/m <sup>2</sup> IV, over 3 hours | days 1-6 |
| • | Crenolanib | 100 mg TID p.o. | starting day 7 (+3 day) |

# Arm B (MEC + crenolanib)

Patients > 18 years of age:

| • | Mitoxantrone | 8 mg/m <sup>2</sup> IV, push | days 1-5 |
|---|--------------|-----------------------------------------|----------|
| • | Etoposide | $100 \text{ mg/m}^2 \text{ IV}$ | days 1-5 |
| • | Cytarabine | 1000 mg/m <sup>2</sup> IV, over 3 hours | days 1-5 |

• Crenolanib 100 mg TID starting day 7 (+3 day)

# Arm C (FLAG-Ida + crenolanib):

Patients > 18 years of age:

| • | Fludarabine | $30 \text{ mg/m}^2 \text{ IV}$ | day 1-5 |
|---|---|---|---|
| • | Cytarabine | 2 g/m <sup>2</sup> IV over 2 hrs | day 1-5 |
| • | G-CSF | 300 ug s.c. inj or IV/5ug/kg SC | day 6 - neutrophil recovery |
| • | Idarubicin | 8 mg/m <sup>2</sup> IV over 30 min | day 1-3 |
| • | Crenolanib | 100 mg TID | starting day 7 (+3 day) |

# **Primary Objective**

• To determine the safety, dose limiting toxicities and maximum tolerated dose (or confirm the target dose of 100 mg TID) of crenolanib given sequentially following standard salvage chemotherapy regimens in subjects with refractory/relapsed AML

## **Secondary Objectives**

- To determine the response rate, duration of response, progression-free survival, and overall survival of crenolanib when given sequentially following standard salvage chemotherapy regimens in subjects with refractory/relapsed AML
- To determine the pharmacokinetics of crenolanib when given sequentially following standard salvage chemotherapy regimens in subjects with refractory/relapsed AML

#### **Inclusion Criteria**

- 1. Confirmed diagnosis of AML, including treatment-related secondary AML (except prior MDS) according to World Health Organization (WHO) 2008 classification at treating institution
- 2. Subjects who are refractory\* or who have relapsed\*\* following first line AML therapy with cytarabine/anthracycline based chemotherapy, with or without a tyrosine kinase inhibitor.

\*Refractory to induction therapy is defined as never achieving CR, CRi or CRp (according to International Working Group criteria) after one line of intensive regimen for AML (reinduction, consolidation and/or transplant allowed) including at least one cytarabine containing induction block with a total dose no less than 700mg/m² per cycle and 3 days of an anthracycline with or without a TKI.

or

\*\*First relapse is defined as untreated hematologic relapse (according to International Working Group criteria) after one line of intensive regimen for AML (re-induction, consolidation and/or transplant allowed) including at least one cytarabine containing induction block with a total dose no less than 700mg/m² per cycle and 3 days of an anthracycline with or without a TKI that induced a CR/CRi/CRp. Subjects are allowed to receive induction, consolidation, transplant and/or maintenance prior to achieving their first CR/CRi/CRp.

- 3. Subjects considered eligible for intensive chemotherapy
- 4. ECOG performance status  $\leq 2$
- 5. Age  $\geq$  18 years
- 6. Adequate liver function within 72 hours of enrollment, defined as:
  - Normal total serum bilirubin
  - ALT and AST  $\leq 2.0 \text{ x ULN}$
- 7. Adequate renal function, defined as serum creatinine  $\leq 1.5 \text{x ULN}$
- 8. Women of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 72 hours prior to enrollment

"Woman of childbearing potential" is defined as any woman who has not undergone a hysterectomy and who has had menses at any time in the preceding 24 consecutive months

9. Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control (IUD, tubal ligation, or partner's vasectomy) while on crenolanib and for 3 months following the last dose of crenolanib.

Hormonal contraception alone is not an acceptable method of birth control for the purpose of this trial.

- 10. Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy and must agree to avoid to father a child (while on therapy and for 3 month after the last dose of crenolanib).
- 11. Willing to adhere to protocol specific requirements
- 12. Following receipt of verbal and written information about the study, the subject must provide

signed informed consent before any study related activity is carried out.

13. Clinically significant toxic effects of prior therapy (expect hydroxyurea) resolved to Grade  $\leq 1$  before the start of study.

#### **Exclusion Criteria**

- 1. < 5% blasts in blood or marrow at screening, except if measurable extramedullary AML is confirmed
- 2. Acute promyelocytic leukemia (APL)
- 3. Known clinically active CNS leukemia
- 4. Clinically active or unstable graft-versus-host disease (GvHD) requiring treatment which precludes administration of chemotherapy as defined in this protocol
- 5. Prior anti-leukemia therapy within 14 days of enrollment for classical cytotoxic agents, and within 5x the half-life for other investigational agents
  - Prior use of hydroxyurea or isolated doses of cytarabine for palliation (i.e., control of WBC) are allowed but should be discontinued at least 24 hrs prior to enrollment.
  - Other agents used strictly with palliative intent might be allowed during this period after discussing with principal investigator
- 6. Pre-existing liver disease (e.g. cirrhosis, chronic hepatitis B or C, nonalcoholic steatohepatitis, sclerosing cholangitis)
- 7. Known HIV infection.
- 8. Evidence of ongoing, uncontrolled systemic infection or an uncontrolled local infection requiring therapy at the start of study.
- 9. "Currently active" second malignancy (other than non-melanoma skin cancer, carcinoma in situ of the cervix or prostatic intraepithelial neoplasia within 1 year). Subjects are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within 1 year.
- 10. Concurrent participation in another therapeutic clinical trial.
- 11. Pregnant or breastfeeding women
- 12. Subjects of childbearing potential not willing to use adequate contraception during study and 3 months after last dose of crenolanib
- 13. Subject with uncontrolled cardiac disease including congestive heart failure class III or IV by the NYHA, unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
- 14. Subject with concurrent severe and/or uncontrolled medical or psychiatric conditions that in the opinion of the investigator may impair the participation in the study or the evaluation of safety and/or efficacy
- 15. Inability to give an informed consent

#### **Statistical Methods**

Initially, the study will evaluate DLT and determine the maximum tolerated dose (or confirm the target dose of 100 mg TID) of crenolanib in combination with either HAM (Arm A), MEC (Arm B) or FLAG-Ida (Arm C) chemotherapy. Thereafter, the study will include a dose-expansion cohort.

For each arm, an initial 6 subjects will be enrolled at a crenolanib dose of 100 mg TID and will be evaluated for DLT, as follows:

- The DLT period will be 28 days
  - Assessment of potential hematologic DLTs that started during the DLT period will extend for up to 6 weeks following the start of the event (see definition of hematologic DLT)
- DLT will be defined as any clinically significant adverse event or abnormal laboratory value that

is not related to concomitant medications, co-morbidities or underlying disease (leukemia), and that is not expected for the chemotherapy being used together with crenolanib

The following will be considered to be DLT:

#### Non-hematologic DLT:

- Any grade 3 or 4 non-hematologic toxicity despite optimal supportive care
  - For example, grade 3 or 4 nausea, vomiting, or diarrhea that cannot be controlled with standard antiemetic or antidiarrheal medications used at optimal dose within 72 hours of onset
- Any tumor lysis syndrome

# **Hematologic DLT:**

- Grade ≥ 3 neutropenia and/or thrombocytopenia with a hypocellular bone marrow lasting for 6 weeks or more after the last dose of therapy in the absence of residual leukemia (i.e., with less than 5% blasts)
  - Anemia will not be considered a DLT

For each arm, prior to determining the maximum tolerated dose (or confirming the target dose of 100 mg TID) of crenolanib based on DLT, subjects will be enrolled in a sequential manner such that no more than 6 subjects are within 30 days of starting induction 1 therapy. See Section 12.2.1 for dose de-escalation and stopping rules based on dose-limiting toxicity.

For each arm, following the determination of the maximum tolerated dose (or the target dose) of crenolanib, subject safety and early mortality will be monitored in cohorts of six throughout the study. Enrollment may be halted at any time based on safety reviews. See Section 12.2.2 for the study's stopping rules following the determination of the maximum tolerated dose (or the target dose) for crenolanib.

Descriptive statistics will be used to summarize the safety and efficacy data for this study. Categorical data will be summarized by number and percentage of subjects in each category. Time-to-event endpoints will be summarized using the cumulative incidence and Kaplan-Meier methodology.

#### 2. BACKGROUND AND STUDY RATIONALE

# 2.1 Unmet Medical Need in Relapsed or Refractory Acute Myeloid Leukemia

Treatment of newly-diagnosed acute myeloid leukemia (AML) with standard chemotherapy regimens, such as anthracyclines and cytarabine, can lead to high complete remission (CR) rates (ranging from 60-70%). Unfortunately, the majority of these patients will relapse. Upon relapse, the prognosis for a second remission or response in these patients significantly worsens.

Currently, there are multiple commonly used AML salvage regimens: high-dose cytarabine, multi-agent chemotherapy, hypomethylating agents, hydroxyurea, and supportive care. Roboz, et al conducted a large international, randomized Phase III clinical trial to investigate the efficacy of elacytarabine (a novel elaidic acid ester of cytarabine) versus investigator's choice of currently available salvage therapies. A total of 381 patients with relapsed/refractory (R/R) AML were enrolled in North America, Europe, and Australia.

The study results showed no significant differences in OS (3.5 v 3.3 months), response rate (23% v 21%), or relapse-free survival (RFS) (5.1 v 3.7 months) between the elacytarabine and control arms, respectively. As shown in Figure 1, overall survival (OS) in both study arms and for all treatments was extremely poor. [36] These results bring to light the need for new treatment options in this patient population.

Figure 1 Overall survival estimates in the intention-to-treat population of elacytarabine versus investigator's choice of current salvage therapies by Kaplan-Meier test



Table 1 30-day, 60-day mortality rates of elacytarabine and investigator's choice

| | Total ITT Population (N=381) | |
|-----------------------|------------------------------|----|
| Parameter | No. of patients | % |
| Early mortality, days | | |
| 30 | 59 | 16 |
| 60 | 117 | 32 |

# 2.2 Physician's Choice of Salvage Chemotherapy Agents in Relapsed/Refractory AML

As mentioned above in section 2.1, Roboz et al showed that there is not a significant difference in OS, RR, or RFS between the elacytarabine and control arm of investigator's choice salvage regimen. Furthermore, figure below, shows the overall survival curves of different salvage regimens (including FLAG-Ida and MEC). These curves show the similarity of the effects of the different salvage regimens on overall survival. MEC and FLAG-Ida had 30 day mortality rates of 19% and 11% respectively. As these salvage regimens have shown similar outcomes, physician's choice of salvage regimen allows the treatment to be chosen based on the individual patient and disease characteristics/status.

Figure 2 Overall survival in the intention-to-treat population of investigator's choice of current salvage therapies by Kaplan-Meier test



## 2.3 Efficacy of HAM, MEC and FLAG-Ida in Relapsed/Refractory AML

MEC and FLAG-Ida have both been shown to provide responses in refractory or early relapse AML patients. In a single-center study, the combination of mitoxantrone, etoposide, and cytarabine (MEC) given as first salvage has shown to achieve a CR of 18% in 77 patients (median age: 54) who were refractory to conventional induction therapy or relapsed after achieving first CR [43]. The efficacy of FLAG-IDA was evaluated as first or second salvage in primary refractory or relapsed AML patients, and a CR/CRi of 73% was reported in 48 patients (median age: 50) [42].

High-dose cytarabine in combination with mitoxantrone (HAM) has also been shown to improve the outcome in patients with R/R AML. Results from a Phase I/II study conducted by the German AML Cooperative Group showed that HAM has high antileukemic activity in refractory AML. High-dose cytarabine with mitoxantrone was associated with a longer OS in patients with poor prognostic features. Of the 40 patients with refractory AML, 21 achieved a complete remission (53%) and 1 patient had a partial remission. [32]

Furthermore, in 2 prospective randomized studies, the high-dose cytarabine with mitoxantrone (HAM) regimen showed significant clinical activity in R/R AML patients (Table 2). In a

prospective randomized pivotal trial, Karanes C et al compared HiDAC (high-dose cytarabine) versus HiDAC + MTZ (mitoxantrone) in relapsed/refractory AML patients. 162 patients were evaluable for response to induction therapy, with 81 patients on each arm. There was trend toward a higher CR rate (from 32% to 44%) with combination HiDAC + MTZ compared to single agent HiDAC. [40]

Kern W et al. performed a randomized study comparing high-dose versus intermediate-dose cytarabine with mitoxantrone in patients with R/R AML. The remission rate and disease free survival were similar in patients getting 3 g/m² of cytarabine for 8 doses as compared to patients getting 1 g/m² of cytarabine for 8 doses. These data suggest that cytarabine at cumulative doses of 6-8 g/m² in combination with MTZ may provide effective complete remission rates in relapsed AML. [31] Hence, this pilot study is using cytarabine at a dose of 6 g/m² along with MTZ as salvage chemotherapy in patients with relapsed AML.

Table 2 Pivotal studies using the HAM regimen as salvage

| Reference | Study design | Regimens | Number of patients | Refractory/<br>relapsed | Median age<br>(yrs) | % CR |
|---|---|---|---|---|---|---|
| Karanes C, et al. 1999 [40] | Phase 3, randomized | HiDAC vs<br>HiDAC +<br>MTZ | 162 (81 on each arm) | 56/106 | 48 vs 53 | 32 vs 44 |
| Kern W, et al.<br>1998 [31] | Phase 3, randomized | HiDAC +<br>MTZ vs<br>IDAC + MTZ | 186 | 27/159 | 50 | 47 |

# 2.4 Clinical Evidence of Combining a Tyrosine Kinase Inhibitor with Chemotherapy in AML Patients

Röllig, et al performed a randomized study (SORAML trial) of sorafenib versus placebo as addon to standard induction in AML patients (irrespective of the Fms-like tyrosine kinase 3 (FLT3) mutation status). Two cycles of induction were allowed (initially with daunorubicin plus cytarabine; patients without response after 1 cycle received a 2<sup>nd</sup> induction with HAM). Consolidation treatment consisted of up to 3 cycles of high-dose cytarabine. 267 patients were enrolled on the study (134 patients received sorafenib and 133 received placebo). Only 46 of 267 (17%) were FLT3 internal tandem duplication (ITD) positive. [34]

Addition of sorafenib to cytarabine/anthracycline chemotherapy resulted in a statistically significant improvement in event-free survival (EFS) (the median EFS was 20.5 months in the sorafenib arm vs. 9.2 months in the placebo arm, p=0.013). These data suggest that in AML patients, the addition of a tyrosine kinase inhibitor (TKI) to standard chemotherapy in a sequential manner is feasible and associated with anti-leukemic efficacy in both FLT3 wild-type and FLT3 ITD AML patients. [34]

Figure 3 Event-free survival in the sorafenib arm vs. placebo



# 2.5 FLT3 Ligand Levels Increase Following Administration of Chemotherapy

It has been shown that plasma FLT3 ligand levels increase by 2-3 log order following intensive chemotherapy in patients with AML. In newly diagnosed AML patients, FLT3 ligand levels rose to 488 pg/mL after course one of chemotherapy and as high as 3251 pg/mL after the fourth course of chemotherapy. [35] These data suggest that the high level of FLT3 ligand in patients following intensive chemotherapy may actually be protective, or even stimulatory, to residual stem cells. Thus, it may be beneficial to add a selective FLT3 inhibitor following chemotherapy.

Figure 4 FLT3 ligand levels increase following multiple regimens of intensive chemotherapy

